CLINICAL TRIAL: NCT05849376
Title: A Pilot Investigation of Emergent Multi-Class Imitation Training (EMIT)
Brief Title: Emergent Multi-Class Imitation Training
Acronym: EMIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Meghan A. Deshais, Ph.D., BCBA-D, Assistant Professor, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro2022001609
Record Dates: First submitted 2023-04-05; First posted 2023-05-08 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism; Imitation
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Intervention Model Description: Single case experimental designs will be used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EMIT Intervention (Experimental): Participants will receive the EMIT intervention.
  Interventions: Behavioral: Emergent Multi-Class Imitation Training

INTERVENTIONS:
Behavioral: Emergent Multi-Class Imitation Training — Sessions will be conducted in a room with minimal distractions containing a table, two chairs, a timer, and 3-4 highly preferred (HP) items identified by preference assessments. A maximum of 10 sessions per week will be distributed across at least 3 days per week. Each session will take 15-20 min to conduct. Novel probe trials will be embedded throughout all sessions to continuously assess for the emergence of generalized imitation. When participants can consistently imitate novel probe responses, the intervention will conclude.

SUMMARY:
The goals of this project are to (a) incorporate empirical findings on imitation training and learning in autistic children into a comprehensive protocol for Applied Behavior Analysis practitioners designed to rapidly facilitate generalized imitation called Emergent Multi-Class Imitation Training (EMIT), and (b) collect pilot data on the efficacy of EMIT with a small sample of autistic children. EMIT will incorporate several features that are grounded in prior research including: (a) evidence-based procedures for establishing trained matching relations (a pre-requisite to generalized imitation), (b) concurrent training of different response types (e.g., motor imitation, object imitation, vocal imitation) to address restricted generalization, (c) multiple manipulative object imitation training, (d) evidence-based procedures for remediating slow acquisition, and (e) frequent tests for the emergence of generalized imitation. EMIT will be the first protocol designed for clinical use that reflects research findings on imitation learning spanning almost five decades.

DETAILED DESCRIPTION:
Using findings from prior research, the investigators will design a manualized training protocol (EMIT) for establishing generalized imitation in autistic children that supervised behavior therapists can implement with a high degree of fidelity. The EMIT protocol will serve as a guide for behavior therapists to help them deliver high-quality, empirically derived imitation training to autistic children. The investigators will conduct a small pilot study to evaluate the effects of EMIT on the emergence of generalized imitation with young autistic children. Single-case experimental design will be used. A multiple baseline across participants design is a single-case design that is common in imitation research with this population. In short, the start of the intervention is stagged across participants to systematically assess the effects of the intervention on each participant's behavior. In this experiment, confirmation that EMIT is responsible for any observed effects will be obtained when changes in each participant's behavior (i.e., correct imitation of novel responses) occur when, and only when, the intervention is introduced.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of autism spectrum disorder
* Age 5 or under
* Maximum score of 40 on Motor Vocal Imitation Assessment
* Demonstrates identity matching above chance levels

Exclusion Criteria:

* Diagnosis of intellectual disability
* Diagnosis of certain conditions that impact motor function (e.g., cerebral palsy)
* Visual impairment
* Hearing impairment

Ages: 12 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Estimated)
Dates: Start 2022-03-27 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Probe performance | Approximately 3x per week throughout participant's EMIT intervention, approximately 3-6 months
  Correct responding to probe trials (novel targets)

SECONDARY OUTCOMES:
Motor Vocal Imitation Assessment | Pre-Intervention and Post-Intervention (within 2 weeks of intervention completion)
  Performance on Motor Vocal Imitation Assessment

CONTACTS AND LOCATIONS:
Overall Officials: Meghan A Deshais, Ph.D., Principal Investigator — Rutgers University
Locations (1):
- Rutgers University, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-12-06): https://cdn.clinicaltrials.gov/large-docs/76/NCT05849376/ICF_000.pdf